CLINICAL TRIAL: NCT05859373
Title: A Randomized, Open Label, Parallel Controlled, Multicenter Phase Ib/II Clinical Trial to Evaluate the Efficacy and Safety of TQB3728 Tablets in Sequential Maintenance of TQB2450 Injection Therapy in Patients After Sequential or Concurrent Chemoradiation for Locally Advanced Non-small Cell Lung Cancer.
Brief Title: To Evaluate the Efficacy and Safety of TQB3728 Tablets in Sequential Maintenance of TQB2450 Injection Therapy in Patients After Sequential or Concurrent Chemoradiation for Locally Advanced Non-small Cell Lung Cancer.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB3728-Ib/II-02
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB3728 tablets+chemoradiation, sequential maintenance with TQB2450 injection (Experimental): TQB3728 tablets combined with sequential or concurrent chemoradiation, 21 days as a treatment cycle. After 4~6 cycles, sequential maintenance therapy of TQB2450 injection.
  Interventions: Combination Product: TQB3728 tablets, TQB2450 injection, sequential or concurrent chemoradiation
- TQB3728 tablets+chemoradiation, sequential maintenance with TQB3728 tablets and TQB2450 injection (Experimental): TQB3728 tablets combined with sequential or concurrent chemoradiation, 21 days as a treatment cycle. After 4~6 cycles, sequential maintenance with TQB3728 tablets and TQB2450 injection for 4 cycles. Then sequential maintenance with TQB2450 injection monotherapy；
  Interventions: Combination Product: TQB3728 tablets, TQB2450 injection, sequential or concurrent chemoradiation
- Sequential or concurrent chemoradiation, sequential maintenance with TQB2450 injection. (Active Comparator): Sequential or concurrent chemoradiation, 21 days as a treatment cycle. After 4~6 cycles, sequential maintenance with TQB2450 injection；
  Interventions: Combination Product: TQB2450 injection, sequential or concurrent chemoradiation

INTERVENTIONS:
Combination Product: TQB3728 tablets, TQB2450 injection, sequential or concurrent chemoradiation — TQB3728 is an inhibitor of apoptosis protein. TQB2450 injection is humanized monoclonal antibody to Programmed Cell Death Protein 1 (PD-1).
  Arms: TQB3728 tablets+chemoradiation, sequential maintenance with TQB2450 injection
Combination Product: TQB3728 tablets, TQB2450 injection, sequential or concurrent chemoradiation — TQB3728 is an inhibitor of apoptosis protein. TQB2450 injection is humanized monoclonal antibody to Programmed Cell Death Protein 1 (PD-1).
  Arms: TQB3728 tablets+chemoradiation, sequential maintenance with TQB3728 tablets and TQB2450 injection
Combination Product: TQB2450 injection, sequential or concurrent chemoradiation — TQB2450 injection is humanized monoclonal antibody to Programmed Cell Death Protein 1 (PD-1).
  Arms: Sequential or concurrent chemoradiation, sequential maintenance with TQB2450 injection.

SUMMARY:
It's a Phase Ib/II clinical trial to evaluate the efficacy and safety of TQB3728 tablets in sequential maintenance TQB2450 injection therapy in patients after sequential or concurrent chemoradiation for locally advanced non-small cell lung cancer.

Incidence and severity of adverse events (AEs), the type of dose-limiting toxicity(ies) (DLT[s]) and Recommended phaseII dose(RP2D) were the Phase Ib primary endpoint. Overall response rate (ORR) was the Phase II primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75 years (calculated based on the date of signing Informed consent form (ICF) ); male or female;
* Non resectable stage III non-small cell lung cancer (NSCLC) patients confirmed by histopathological or cytological examination；
* At least one measurable lesion (based on RECIST 1.1)；
* Has not received any systematic treatment or targeted radiotherapy for locally advanced non-small cell lung cancer;
* Eastern cooperative oncology group (ECOG) score 0-1;
* Estimated survival time ≥ 3 months;
* The main organs function are normally, meeting following criteria:

  1. routine blood tests: hemoglobin (HGB) ≥80g/L (no blood transfusion and blood products within 14 days); absolute neutrophil count (ANC) ≥1.5×109/L; platelets (PLT)≥90×10^9/L.
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN);Serum creatinine (CR) ≤ 1.5×ULN or creatinine clearance (CCR) ≥ 60 ml/min.
  3. Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy);
  4. Cardiac ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%.
* Female participants should have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Participants should agree that contraception must be used during the study period and for 6 months after the end of the study.

Exclusion Criteria:

* Comorbidity and medical history:

  1. Have had or currently have other malignant tumors within 2 years. The following two conditions can be enrolled: other malignancies treated with a single surgery; cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumors), Tis (carcinoma in situ) and T1 (tumor-invasive basement membrane)];
  2. Pathological types of mixed small cell and non-small cell lung cancer components；
  3. Patients with known EGFR/ALK mutations
  4. There was Therapeutic toxicity (≥ CTC AE grade 2 infection)
  5. Have a history of idiopathic pulmonary fibrosis, organized pneumonia, drug-induced pneumonia, or idiopathic pneumonia
  6. Subjects who have received major surgical treatment or obvious traumatic injury within 4 weeks prior to initial administration
* Tumor related symptoms and treatment

  1. Received Antitumor traditional Chinese medicine treatment within 2 weeks before the start of research treatment；
  2. Previously received other PD-1/PD-L1/CTLA-4 antibody treatments or immunotherapy;
  3. Uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage;
* Research treatment related:

  1. Subjects who have received the vaccine within 4 weeks prior to the first dose, or is planning to be vaccinated during the study period
  2. Individuals with a previous history of severe allergies to macromolecular drugs or severe hypersensitivity reactions after administration of other monoclonal antibodies
  3. Existence of any active autoimmune disease or history of autoimmune disease
* Subjects who have participated in clinical trials of other anti-tumor drugs within 4 weeks before the first dose
* According to the judgment of the investigator, subjects with concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects with other reasons which are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Baseline to 30 days after last administration.
  All adverse medical events that occur after the subject receives the investigational drug evaluated according to the National Cancer Institute standard for common toxic reactions (NCI-CTC) V5.0.
Severity of adverse events (AEs) | Baseline to 30 days after last administration.
  All adverse medical events that occur after the subject receives the investigational drug evaluated according to the National Cancer Institute standard for common toxic reactions (NCI-CTC) V5.0.
Dose-limiting toxicity (DLT) | Up to 28 days.
  Subjects within 28 days after treatment appear the following toxicity reaction relate to the drug: grade III or above of non-hematological toxicity, grade IV hematological toxicity, neutropenia associated with fever.
Recommended phase II dose (RP2D) | Baseline to 30 days after last administration.
  The RP2D defined as the lower dose level to maximum tolerated dose based on the safety profile.
Overall response rate (ORR) | Baseline to the disease progression, up to two years.
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, the proportion of subjects whose tumors are evaluated as complete response (CR) and partial response (PR) by subcenter imaging evaluation. It is recorded from the first dose of the drug to disease progression or initiation of a new anticancer treatment.

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (Tmax) | For single dose, pre-dose, 0.5,1, 2, 3, 4, 8, 24 hours after dose; For multiple dose, pre-dose on day 3, day 5, day 7, day 14 and 0.5, 1, 2, 4, 8, 24, 48, 72 hours after dose on day14.
  To characterize the pharmacokinetics of TQB3728 by assessment of time to reach maximum plasma concentration.
Peak concentration (Cmax) | For single dose, pre-dose, 0.5,1, 2, 3, 4, 8, 24 hours after dose; For multiple dose, pre-dose on day 3, day 5, day 7, day 14 and 0.5, 1, 2, 4, 8, 24, 48, 72 hours after dose on day14.
  Cmax is the maximum plasma concentration of TQB3728 or metabolite(s).
Terminal half-life (t1/2) | For single dose, pre-dose, 0.5,1, 2, 3, 4, 8, 24 hours after dose; For multiple dose, pre-dose on day 3, day 5, day 7, day 14 and 0.5, 1, 2, 4, 8, 24, 48, 72 hours after dose on day14.
  Pharmacokinetics parameters to evaluate the half life of TQB3728.
Area under the plasma concentration-time curve from time zero to time t. | For single dose, pre-dose, 0.5,1, 2, 3, 4, 8, 24 hours after dose; For multiple dose, pre-dose on day 3, day 5, day 7, day 14 and 0.5, 1, 2, 4, 8, 24, 48, 72 hours after dose on day14.
  To characterize the pharmacokinetics of TQB3728 by assessment of area under the plasma concentration time curve from zero to specific time or infinity.
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) | For single dose, pre-dose, 0.5,1, 2, 3, 4, 8, 24 hours after dose; For multiple dose, pre-dose on day 3, day 5, day 7, day 14 and 0.5, 1, 2, 4, 8, 24, 48, 72 hours after dose on day14.
  Cmax,ss is the steady state maximum concentration of TQB3728.
Minimum steady-state plasma drug concentration during a dosage interval (Cmin,ss) | For single dose, pre-dose, 0.5,1, 2, 3, 4, 8, 24 hours after dose; For multiple dose, pre-dose on day 3, day 5, day 7, day 14 and 0.5, 1, 2, 4, 8, 24, 48, 72 hours after dose on day14.
  Cmin,ss is the minimum plasma concentration of TQB3728.
Disease control rate (DCR) | Baseline to up to two years.
  Percentage of subjects achieving CR and PR and stable disease (SD).
Duration of Response (DOR) | Baseline to up to two years.
  The period from the subjects first achieving CR or PR to disease progression.
Progression-free survival (PFS) at 12 months. | Up to 12 months.
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Progression-free survival at 18 months. | Up to 18 months.
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Progression-free survival. | Baseline to the disease progression, up to two years.
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) at 12 months. | Up to 12 months.
  OS is defined as the time from the first administration to all-cause death.
Overall survival (OS) at 18 months. | Up to 18 months.
  OS is defined as the time from the first administration to all-cause death.
Overall survival (OS) | Baseline to the disease progression, up to two years.
  OS is defined as the time from the first administration to all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China